CLINICAL TRIAL: NCT03060889
Title: Tranexamic Acid Use in Elective Cesarean Section for Women With Placenta Previa: A Randomized Controlled Trial
Brief Title: Tranexamic Acid Use in Elective Cesarean Section for Women With Placenta Previa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed Hassan Elbohoty, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAbdelaziz
Record Dates: First submitted 2017-01-10; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Placenta Previa
Keywords: Cesarean section; placenta previa; Tranexamic acid
MeSH Terms: conditions — Placenta Previa | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cases (Active Comparator): Tranexamic acid 10 mg/ kg body weight will be given by intravenous infusion with induction of anesthesia in elective cesarean section for non complicated cases of placenta previa
  Interventions: Drug: Tranexamic acid
- Controls (No Intervention): Control group will not receive Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — 10 mg/kg body weight will be given with induction of anesthesia by intravenous infusion
  Arms: Cases

SUMMARY:
Tranexamic Acid Use in Elective Cesarean Section for Women With Placenta Previa

DETAILED DESCRIPTION:
Tranexamic Acid Use in Elective Cesarean Section for Women With Placenta Previa to detect efficacy of Tranexamic acid in decreasing blood loss

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy (more than 37 weeks of gestation)
* Diagnosis of placenta previa was confirmed by ultrasound
* The patient hemoglobin percentage is more than 10 mg/dl

Exclusion Criteria:

* Invading placenta previa diagnosis was confirmed by Doppler ultrasound studies
* Emergency lower segment cesarean section
* Associated medical comorbidities

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-02; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
intra operative blood loss in ml | intraoperative during cesarean section
  Calculation of blood loss during cesarean section in the two groups to detect efficacy of Tranexamic acid in reducing blood loss

IPD SHARING:
Plan to Share IPD: Undecided